CLINICAL TRIAL: NCT02102321
Title: A Randomized Effectiveness Trial of Hookworm Treatment of Women Smallholder Farmers to Evaluate Improved Productivity of Their Farming and/or Household Labor
Brief Title: Does Treating Hookworm Improve Productivity of Small Subsistence Farmers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salmon, Margaret, M.D. (Individual)
Collaborators: Akeso Associates (Unknown); Bill and Melinda Gates Foundation (Other); Eastern Congo Initiative (Unknown); HEAL Hospital, DRC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HW0001
Record Dates: First submitted 2014-03-29; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Hookworm Stool Burden; Anemia; Exercise Tolerance
Keywords: hookworm; albendazole; iron supplementation; democratic republic of congo; subsistence farmers; randomized control trial; neglected tropical disease; helminths
MeSH Terms: conditions — Anemia; Ancylostomiasis; Neglected Diseases | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- albendazole (Experimental): albendazole 400 mg
  Interventions: Drug: albendazole
- placebo (Active Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: albendazole
  Arms: albendazole
Drug: placebo
  Arms: placebo

SUMMARY:
Treatment of hookworm infected groups with albendazole has been shown to result in an increase in hemoglobin levels and a related decrease in the prevalence of anemia. Increases in hemoglobin levels due to treatment have been associated with significant gains in adult labor productivity.

In this study, the investigators hypothesize that regular treatment of women smallholder farmers in a high prevalence area with the anti-hookworm drug albendazole and iron supplementation will improve hookworm associated anemia. Further, regular treatment of albendazole and iron supplementation will improve their work capacity when compared to a control group

DETAILED DESCRIPTION:
DRC has one of the world's highest prevalences (frequencies) of Soil Transmitted Helminths (STH), a group of intestinal parasites that include Ascaris, Trichuris and hookworm, each of which can have significant impacts on the health and nutritional status of children.(1)(2)(3) In addition, hookworm, because of prevalence increases noted during adulthood in many countries and because of its relationship to significant intestinal blood loss, can also have a significant impact on the health and nutritional status of adults.

Hookworm spreads easily in places without adequate control of feces; hookworm eggs are excreted in feces of infected people, transition to larvae, and usually enter the body through the skin on the bottom of the feet of other people who are not wearing footwear.

Much of hookworm's health impact is mediated through intestinal blood loss as hookworms attach to the human intestinal wall and digest the hemoglobin in human red blood cells. That blood loss leads to - or exacerbates - iron deficiency and eventually to iron deficiency anemia (IDA). Because of menstrual blood losses, the large iron demands of pregnancy, and the often low iron content of their diets, many women of childbearing age are at risk of iron deficiency even without hookworm exposure. Any blood loss associated with hookworm infection would exacerbate a pre-existing iron deficiency.

Iron deficiency with or without anemia has also been associated in several studies with lower aerobic work capacity. IDA can effect an individual's ability to perform economic generating tasks (work output) threaten one's livelihood and possibly food security. The World Health Organization (WHO) estimates an annual loss of 19.7 million disability-adjusted life years (1.3% of the global total) is due to IDA with high burden in Africa (25%), an area which can least afford it. The median annual economic loss due to IDA has been estimated at 4% of gross domestic product in 10 different developing countries.

Albendazole and Mebendazole are anti-helminthic drugs that that can cure or reduce the severity (as measured by stool egg counts) of many hookworm infections. The major programmatic use of these drugs is in programs of school-based mass drug administration (MDA) as recommended treatment strategies have traditionally prioritized school-aged children. Large amounts of these drugs are now being provided without charge by their manufacturers, Merck and Johnson & Johnson respectively, and distributed through W.H.O. and ministries of health to support current goals of control of pediatric hookworm and other STH infections.

Treatment of hookworm infected groups with Albendazole has been shown to result in an increase in hemoglobin levels and a related decrease in the prevalence of anemia. Increases in hemoglobin levels due to treatment have also been associated with significant gains in adult labor productivity as measured in Kenyan road construction workers (16) and in Bangladeshi women plantation tea pickers. However, the cure or amelioration of hookworm infection caused by these drugs is not permanent; re-infection can occur within weeks or months in heavily exposed people. Few studies have measured work productivity beyond 2-3 months and minimal information is available for longer term treatment.

This study is in response to the Bill and Melinda Gates Foundation Grand Challenges Explorations RFP targeted specifically at "Labor Saving Strategies and Innovations for Women Smallholder Farmers." As hookworm in endemic areas is thought to be one of the primary causes of IDA and IDA is known to decrease work productivity, then subsistence farmers will ideally report improved productivity if hookworm is treated. Although the benefits of this proposed intervention are not directly targeted at that specific goal, i.e., are not intended to reduce the amount of necessary labor, the benefits of this intervention could lead indirectly to the same result(s) through an increase of women's ability to accomplish a fixed amount of work.

The Democratic Republic of Congo is thought to be an appropriate location as it has one of the world's highest burdens of NTD disease with an estimated 31 million hookworm cases, second only to Nigeria for disease prevalence in Africa. The population is also particularly vulnerable as moderate to heavy hookworm infections has been associated with lower hemoglobin levels (in both children and adults) and thus with a greater risk of iron deficiency and anemia. DRC has also been identified by USAID as a country in need of urgent NTD disease surveillance and control activities. Information from this study will ideally extend understanding of this disease process and provide information regarding inclusion of anthelmintic treatment in maternal and other public health packages.

Study Purpose The purpose of this study is to determine whether regular treatment of women smallholder farmers with the anti-hookworm drug Albendazole over a one-year period would have an impact on their work capacity and possible productivity as small farmers. The intention is to identify and enroll in an intervention study a group of women smallholder farmers who are not pregnant in their first trimester of pregnancy, are not acutely ill with malaria, and living in areas with poor sanitation and with endemic hookworm. Many of these women would presumably be iron deficient, at least in part due to the blood loss associated with hookworm infection.

Study Aims

1. To determine prevalence of hookworm infection in the Safe Motherhood cohort
2. To determine the prevalence of anemia in the Safe Motherhood cohort
3. To determine the change in Hemoglobin of female subsistence small farmers who have been treated with Albendazole and daily iron supplementation at 6 and 12 months.
4. To determine the change in work tolerance as measured by the STEP test when female subsistence small farmers have been given Albenzazole and iron supplementation at 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* All women of childbearing years (age 16 - 50)
* Identify as a small subsistence farmer
* No clinical evidence of acute malaria, who are with hookworm + stool, and are not pregnant.

If women become pregnant during the period of study and tests + at the 6 or 12 month study visit then based on last menstrual period, we will wait until she has completed her first trimester to initiate the 6 or 12 month study visit based on protocol.

Exclusion Criteria:

* Women with acute symptoms of malaria
* 1st trimester pregnancy
* Hookworm - stool
* Declines study participation
* Age <16 or > 50
* Muscular or neurologic defect that preclude them from stepping on and off a stairs
* Cognitive impairment such that they cannot understand study purpose and consenting procedure

Ages: 17 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Exercise Tolerance Harvard STEP Test | 12 months
  Subjects exercise tolerance will be measured as amount of time able to step on and off the Harvard Step and the heart rate as measured in beats per minute after a 5 minute step interval

SECONDARY OUTCOMES:
albendazole efficacy | 12 months
  subjects stool will be retested for hookworm burden at 14 days and 3 months after treatment with albendazole to determine the percentage treatment failure rate.
hemoglobin | 12 months
  Subjects hemoglobin will be measured at study start, at 6 months and at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Salmon, MD MPH, Principal Investigator — University Health Network, Toronto; Christian Salmon, DrSc, Principal Investigator — Western New England University
Locations (1):
- Safe Motherhood Cohort, Idgwi Island, South Kivu, Republic of the Congo